CLINICAL TRIAL: NCT04823195
Title: Development of Cellular Models of the Ear and Nose From Patient Samples to Study the Mechanisms of Hearing
Brief Title: Development Cellular Models of the Ear and Nose to Study the Mechanisms of Hearing
Acronym: CMAG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0331
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Hearing Loss, GJB2, Cis Regulation, DFNB1
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Development of cells culturesissued from Nose and Ear to study auditory mecanisms.

Study of the cis-Modulation of the gene GJB2 for the patients with early presbycusis to identify the genetic cause of hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Hearing loss Presbycusis Exostosis

Exclusion Criteria:

* Genetic hearing loss

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: over 18 years old full consent With exostosis, or having cochlear implant surgery, or early presbycusis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
GJB2 cis regulation | 2 years
  Culture cell model

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning two years and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.